CLINICAL TRIAL: NCT00975091
Title: A Study of the Safety and Antiviral Activity of Open-Label Entecavir (BMS-200475) in Adults With Chronic Hepatitis B Infection Who Have Completed Dosing in a Previous Phase II/III Study in China
Brief Title: Continue Entecavir Rollover From China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI463-050
Record Dates: First submitted 2009-09-08; First posted 2009-09-11 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entecavir 0.5 (Active Comparator)
  Interventions: Drug: Entecavir
- Entecavir 1.0 (Active Comparator)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 0.5 mg, once daily, Until ETV is commercially available in China or when Post Study Drug Program is started
  Other Names: Baraclude; BMS-200475
  Arms: Entecavir 0.5
Drug: Entecavir — Tablets, Oral, 1.0 mg, once daily, Until ETV is commercially available in China or when Post Study Drug Program is started
  Other Names: Baraclude; BMS-200475
  Arms: Entecavir 1.0

SUMMARY:
The purpose of the study is to determine if treatment with entecavir is safe and well tolerated in patients who completed dosing in a previous entecavir study in China, but are requiring further treatment of their chronic hepatitis B virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had completed the required dosing period in a previous ETV Phase 2 or 3 study in China (studies AI463012, AI463023, AI463056), and had been assessed by the Investigators as likely to benefit from additional therapy for treatment of their HBV infection
* ALT ≤ 15 x upper limit of normal
* Compensated liver disease

Exclusion Criteria:

* Coinfection with HIV, HCV, or HDV

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2004-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The number and percentage of subjects with adverse events, laboratory abnormalities, and discontinuations due to adverse events | Through 3 years of dosing and up to 48 weeks of off treatment follow up

SECONDARY OUTCOMES:
The change in the mean HBV DNA measured by PCR assay from baseline for each entecavir cohort | Through 3 years of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb